CLINICAL TRIAL: NCT04220463
Title: HYVIR : Interest of Hypnosis During the Implementation of Non-invasive Ventilation in a Patient With COPD and/or Obesity With a BMI Greater Than 30, Conscious With Acute Respiratory Distress in the Adult Intensive Care Unit
Brief Title: Interest of Hypnosis When Setting up Non-invasive Ventilation in a Conscious Patient With COPD and/or Obesity With a BMI Greater Than 30, Suffering Fromacute Respiratory Distress in Adult Intensive Care
Acronym: HYVIR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 35RC19_9747_HYVIR; 2019-A02238-49 (Other: ID RCB); 19/08/14/42258 (Other: CNRIPH)
Record Dates: First submitted 2019-12-20; First posted 2020-01-07 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Obesity With a BMI Greater Than 30; Acute Respiratory Distress in Adult Intensive Care
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Hypnosis; Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: Prospective monocentric, controlled, randomized, superiority, open study with a blind assessor, on two parallel groups.
Who Masked: Outcomes Assessor
Masking Description: Patient randomization will be done online.
  SETTING UP AND MAINTAINING THE INSU People having knowledge of the randomization group
  * Doctor in charge of the patient
  * Doctor/IDE dedicated to hypnosis (present throughout the procedure, regardless of the randomization group)
  * Patient People not having knowledge of the randomization group
  * assessor = other IDE or doctor not directly taking care of the patient assessor present at 4 times: inclusion, H0, H2 and H24 but absent during the procedure 1 single assessor for the 4 times of the same patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnosis group (Experimental): For the hypnosis group, hypnotic support is set up by a doctor/IDE previously trained and dedicated during the implementation of the NIV. The dedicated doctor/IDE will be presented before the start of the NIV setup procedure and will start the hypnosis session a few minutes before the mask is put on. The procedure for setting up the NAV may begin after agreement from the dedicated doctor/IDE.
  Interventions: Other: Hypnosis + NIV
- Control group (Placebo Comparator): In the control group, in order to preserve the knowledge of the evaluator, the doctor/IDE dedicated to hypnosis is present in the service but does not intervene in the care so as not to be tempted to involuntarily put hypnosis in place. The assessor will be chosen from the two other teams present in the other two modules (each module is a seven-bed unit and has no physical communication with the other two) after the start of the procedure for setting up the NIV, with or without hypnosis, in order to be certain that he had no visual contact with the patient and the caregivers present before the evaluation. The implementation of the NAV will take place as usually carried out in the service.
  Interventions: Other: NIV

INTERVENTIONS:
Other: Hypnosis + NIV — For the hypnosis group, hypnotic support is set up by a doctor/IDE previously trained and dedicated during the implementation of the NIV. The dedicated doctor/IDE will be presented before the start of the NIV setup procedure and will start the hypnosis session a few minutes before the mask is put on. The procedure for setting up the NAV may begin after agreement from the dedicated doctor/IDE.
  Arms: Hypnosis group
Other: NIV — In the control group, in order to preserve the knowledge of the evaluator, the doctor/IDE dedicated to hypnosis is present in the service but does not intervene in the care so as not to be tempted to involuntarily put hypnosis in place. The assessor will be chosen from the two other teams present in the other two modules (each module is a seven-bed unit and has no physical communication with the other two) after the start of the procedure for setting up the NIV, with or without hypnosis, in order to be certain that he had no visual contact with the patient and the caregivers present before the evaluation. The implementation of the NAV will take place as usually carried out in the service.
  Arms: Control group

SUMMARY:
Discomfort during respiratory decompensation of a patient with chronic obstructive pulmonary disease (COPD) and/or obesity with a BMI greater than 30, in intensive care and the establishment of non-invasive ventilation (NIV) is frequent and a source of failure. this therapy. Pharmacological treatments may be impossible due to the pathology, the risk of it worsening and adverse effects. In this context, hypnosis appears to be a tool that would promote comfort and thus increase tolerance of NIV.

ELIGIBILITY:
Pre-inclusion criteria

* Man or woman, aged 18 or over, admitted to medical intensive care
* Glasgow score = 15
* Patient with acute respiratory failure decompensating COPD and/or having obesity with a body mass index (BMI) greater than 30
* Patient having given free, informed and written consent
* Patient affiliated to a health insurance system

Inclusion Criteria:

* Glasgow score = 15
* Need during use of non-invasive ventilation

Exclusion Criteria:

* Procedure to be carried out in extreme urgency (PaCO2 too high and leading to an immediate vital risk, and / or PaO2 too low) on medical decision
* Confusional state making hypnosis impossible
* Decompensated psychiatric illness
* Patient entering with an NIV in place already installed in another department. The subject becomes included again at the end of the treatment with NIV if however he needs it again.
* Patient already included in the study during previous non-invasive ventilation
* Patient participating in research involving an interventional human person (category 1) on an analgesic / sedative medication
* A person of full age subject to legal protection (safeguard of justice, curators, guardianship) or deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-11-20 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
Comfort | 2 hours after initiation of NIV
  Quantification of comfort by a Digital Verbal Comfort Scale 2 hours after initiation of NIV (from 0 to 10, 0 being the minimum comfort felt and 10 the maximum comfort felt by the patient)

SECONDARY OUTCOMES:
Anxiety | Before and 30 minuts, 2 hours and 24 hours after the implementation of the NIV
  Assessment of anxiety (Numerical Verbal Scale from 0 to 10) at inclusion, 30 minutes, 2 hours and 24 hours after the implementation of the NIV
First NIV session duration | At the end of the first NIV session
  Calculation of the number of hours of the first NIV session
Comfort | Before and 30 minuts and 24 hours after the implementation of the NIV
  Comfort assessment at inclusion, 30 minutes and 24 hours after the implementation of the NIV (Digital Verbal Scale from 0 to 10)
TcpCO2 | Before and 30 minuts, 2 hours and 24 hours after the implementation of the NIV
  Decrease in PaCO2: Installation of a transcutaneous sensor and measurement of TcpCO2 at inclusion, 30 minutes, 2 hours and 24 hours after the establishment of the NIV
NIV duration | after the first 24 hours of treatment
  Calculation of the number of hours of NIV in the first 24 hours of treatment
dyspnea | 2 hours after the setting up of the NIV
  Assessment of the dyspnea felt by the patient 2 hours after the setting up of the NIV: +2: significant improvement; +1 slight improvement; 0 No change; -1 slight deterioration; -2 significant deterioration.
Intubation | Day 28
  Number of intubations: calculation of the number of patients intubated during the ICU stay.
Stay duration | Day 28
  Duration of stay in intensive care
anxiolytic treatment prescription | Day 28
  Record of the number of patients who had to have a prescription for anxiolytics during hospitalization in intensive care.
stress | Before and 30 minuts and 2 hours after the implementation of the NIV
  Evaluation of the stress of the healthcare team by a numerical verbal scale from 0 to 10 (0 being no stress and 10 the greatest possible stress felt) at inclusion, 30 minutes and 2 hours after NIV initiation

CONTACTS AND LOCATIONS:
Locations (1):
- Rennes University Hospital, Rennes, Brittany Region, France

IPD SHARING:
Plan to Share IPD: No